CLINICAL TRIAL: NCT05453695
Title: Intravenous DNase I for the Treatment of Sepsis: A Phase I Safety and Feasibility Study in ICU Patients
Brief Title: Intravenous DNase I for the Treatment of Sepsis (IDEALSepsisI)
Acronym: IDEALSepsisI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDEALSepsisI
Record Dates: First submitted 2022-06-24; First posted 2022-07-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sepsis; Critical Illness
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous DNase I (Experimental): We will enroll up to 36 Participants; each is receiving repeated unit doses of DNase I, BID, delivered by IV infusion over 3 or 7 consecutive days (12 +/- 1 hour apart) according to the following dose-escalation schedule with up to 6 Participants per dose panel.
  * Panel 1: 25 µg/kg, BID for 3 days (cumulative dose: 150 µg/kg)
  * Panel 2: 25 µg/kg, BID for 7 days (cumulative dose: 350 µg/kg)
  * Panel 3: 125 µg/kg, BID for 3 days (cumulative dose: 750 µg/kg)
  * Panel 4: 125 µg/kg, BID for 7 days (cumulative dose: 1750 µg/kg)
  Interventions: Drug: Intravenous DNase I
- Control (No Intervention): We will also enroll 12 septic Participants who do not receive intravenous DNase I (as Comparator Group). These patients will be recruited contemporaneously based on the same inclusion and exclusion criteria.

INTERVENTIONS:
Drug: Intravenous DNase I — Dose-escalating intravenous infusion of DNase I
  Arms: Intravenous DNase I

SUMMARY:
Phase I dose-escalation safety and feasibility of IV DNase I in ICU septic patients.

DETAILED DESCRIPTION:
In sepsis, the release of 'neutrophil extracellular traps' (NETs) by activated neutrophils may contribute to organ damage by acting as scaffolds that trap blood cells and fibrin clots. Excessive NET formation can occlude the vasculature, promoting thrombosis and tissue hypoperfusion. This is a trial on a novel IV therapy for septic patients that shows promise in multiple animal models of sepsis. The therapy, DNase I, is an enzyme that helps to dismantle NETs by digesting cell-free DNA (cfDNA), the major structural component of NETs. The objective of this study is to conduct a Phase I dose-escalation safety and feasibility of IV DNase I in ICU septic patients. The results of this study may justify a future Phase II trial of the efficacy and safety of DNase I for critically ill patients with sepsis.

This trial proposes

1. - To determine the safety, feasibility and maximum tolerated dose (MTD) of using DNase I in septic patients
2. - To evaluate clinical endpoints common in the critically ill such as organ dysfunction severity and trajectory, ICU length of stay, and mortality.
3. - To describe the effects of DNase I on blood coagulation and NETs release
4. - To collect samples for future studies on coagulation and immune function in sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥18 years
2. Admitted to the ICU in the last 48 hours
3. Suspected or proven infection as the admitting diagnosis
4. A sequential (sepsis) organ function assessment (SOFA) score of ≥2 above baseline
5. Expected to remain in the ICU for ≥ 72 hours

Exclusion Criteria:

1. No consent/inability to obtain consent from a substitute decision-maker
2. Have other forms of clinically apparent shock, including cardiogenic, obstructive (massive pulmonary embolism, cardiac tamponade, tension pneumothorax), hemorrhagic, neurogenic, or anaphylactic shock
3. Have a significant risk of bleeding as evidenced by one of the following:

   * Surgery requiring general or spinal anesthesia within 24 hours before enrolment
   * The potential need for surgery in the next 24 hours
   * Evidence of active bleeding
   * A history of severe head trauma requiring hospitalization
   * Intracranial surgery, or stroke within three months before the study
   * Any history of intracerebral arteriovenous malformation, cerebral aneurysm, or mass lesions of the central nervous system
   * A history of congenital bleeding diatheses
   * Gastrointestinal bleeding within five weeks before the study unless corrective surgery had been performed
   * Trauma is considered to increase the risk of bleeding
   * Presence of an epidural catheter
   * Need for therapeutic anticoagulation
4. Receiving DNase I by inhalation
5. Terminal illness with a life expectancy of fewer than three months
6. Pregnant and/or breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients recruited per month from the start of the study | up to 24 months
  Number of patients recruited per month
Number of patients who completed the protocol | up to 7 days
  The ability to complete study infusion and blood collection as prescribed

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score | Baseline to Day 10
  Quantitative variable: Maximal score of SOFA (Sequential Organ Failure Assessment) will be recorded; Value range 0-24 points
  * Delta SOFA score, defined as maximum versus minimum SOFA during ICU stay
  * Change in SOFA score within 48 hours
Organ support free days | at Day 28
  Increase of three or more days free from vasopressor therapy, invasive mechanical ventilation or renal replacement therapy.
Duration of ICU admission | up to 9 months
  Number of days since admission to discharge from the ICU
Time to Hospital discharge | up to 90 days
  Time elapsed between enrolment into the study (at admission), and discharge
Mortality at Day 90 | up to day 90
  Number of patients alive at day 90
European Quality of Life (EuroQol) - 5 Domain 5 Level Scale (EQ-5D-5L) Utility Score | At day 90
  Average or median EQ-5D-5L score
Collection of Research Biomarkers related to inflammation and coagulation | up to day 14
  Number of patients with all sets of biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma N, Dwivedi DJ, Fux L, Hayon Y, Ruderfer I, Nataf Y, Cani E, Liaw PC. Intravenous Delivery of Long-Acting Dnase I (PRX-119) In a Murine Model of Polymicrobial Abdominal Sepsis. Shock. 2026 Jan 1;65(1):76-84. doi: 10.1097/SHK.0000000000002666. Epub 2025 Jul 8. PMID 40705350